CLINICAL TRIAL: NCT02254525
Title: A Multicenter, Randomized, Double-blind, and Parallel Groups, Placebo-controlled Trial of the Efficacy and Safety of a New Formulation of Ibuprofen 800 mg Every 6 Hours in the Management of Postoperative Pain.
Brief Title: A Multicenter Trial of the Efficacy and Safety of a New Formulation of Ibuprofen 800 mg Every 6 Hours in the Management of Postoperative Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sample not reached in traumathology arm
Sponsor: Biomendi S.A.U. (Industry)
Collaborators: Pivotal S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIBEC02
Record Dates: First submitted 2014-09-25; First posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ibuprofen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 800 mg intravenous ibuprofen (Experimental): Treatment group: 800 mg IV ibuprofen, starting at the moment of skin closure and every 6 hours, infused over 15 minutes.
  Interventions: Drug: Intravenous ibuprofen
- 200 ml of saline solution (Placebo Comparator): Placebo group: 200 ml of saline solution, starting at the moment of skin closure and every 6 hours, infused over 15 min.
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: Intravenous ibuprofen — Treatment group: 800 mg IV ibuprofen, starting at the moment of skin closure and every 6 hours up to 72 hours after the first dose.
  All patients will receive morphine administered by patient controlled analgesia (PCA). Investigation treatment will be administered every 6 hours until 24 h in abdominal surgery, 48 h in hip surgery and 72 h in knee surgery.
  Other Names: IV ibuprofen
  Arms: 800 mg intravenous ibuprofen
Drug: Saline solution — Placebo group: 200 ml of saline solution, starting at the moment of skin closure and every 6 hours up to 72 hours after the first dose.
  All patients will receive morphine administered by patient controlled analgesia (PCA). Investigation treatment will be administered every 6 hours until 24 h in abdominal surgery, 48 h in hip surgery and 72 h in knee surgery.
  Other Names: Placebo
  Arms: 200 ml of saline solution

SUMMARY:
The purpose of this study is to study the efficacy of intravenous administration of ibuprofen compared to placebo in patients with postoperative pain and evaluate its tolerability and safety profile.

DETAILED DESCRIPTION:
This is a phase III, national, multicenter, randomized, double-blind, parallel groups, and placebo-controlled.

Patients will be randomized to receive either ibuprofen or placebo. Stratified randomization will be used to assign eligible patients to a stratum according to type of surgery and centre. Randomization sequence will be generated in the coordinating centre.

Blinding of the patient and study personnel evaluating response will be warranted by adequate drug labelling.

All patients will receive morphine administered by patient controlled analgesia (PCA) following a similar schedule in all centres: 1 mg bolus dose with a close time of 5 min and a maximum of 10 mg in an hour and a maximum of 30 mg in 4 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women between 18 and 80 years old.
2. Being scheduled for elective single surgical site orthopaedic surgery (hip or knee joint replacement, corsed ligaments, column or shoulder surgery), or abdominal surgery (inguinal hernia, cholecystectomy, eventration or hiatus hernia)
3. Being scheduled for general anaesthesia or regional anesthesia without regional analgesia after surgery.
4. Having anticipated need for postoperative narcotic analgesia administered by patient controlled analgesia (PCA).
5. Expected to stay at the hospital for at least 24 h.
6. Providing written informed consent for participating in this study.

Exclusion Criteria:

1. Use of NSAID within 12 hours prior to the first planned dose.
2. Taking oral anticoagulants, lithium, combination of ACE inhibitors, furosemide or aspirin.
3. Anaemia (haemoglobin <10 g/dl) and/or history or evidence of asthma or heart failure.
4. History of allergy or hypersensitivity to any component of IV ibuprofen, aspirin or aspirin related products, NSAID or COX-2 inhibitors.
5. Pregnant or nursing.
6. Weight less than 40 kg.
7. History of severe head trauma that required hospitalization, intracranial surgery or stroke within the previous 30 days, or any history of intracerebral arteriovenous malformation, cerebral aneurism or CNS mass lesion.
8. History of congenital bleeding diathesis or any active clinically significant bleeding or underlying platelet dysfunction.
9. Gastrointestinal bleeding that required medical intervention.
10. Platelet count less than 80.000 determined within the 28 days prior to surgery.
11. Pre-existing dependence on narcotics or receiving chronic treatment with opioids.
12. Severe renal failure (calculated creatinine clearance < 60 ml/min).
13. Liver failure, ALAT or ASAT >3 times upper limit of normality, or bilirubin >2 g/dl.
14. Diagnosed of Bowel Inflammatory Disease.
15. Not able to understand the requirements of the study, or to abide by the study restrictions or to return for the required assessments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2012-05; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of intravenous ibuprofen for the management of postoperative pain in comparison to placebo | First 24 hours post- surgery
  The primary efficacy endpoint will be the reduction in total morphine use in the first 24 hours post- surgery as compared to placebo.

SECONDARY OUTCOMES:
Secondary efficacy endpoints | From 0 hours to 72 hours post- surgery
  - Consumption of morphine in the first 48 h (and 72) hours post- surgery.
Secondary efficacy endpoints | From 0 hours to 72 hours post- surgery
  - Pain intensity at rest and with movement measured with the eleven points visual analogue scale (VAS), at 1 and 3 hours and every 6 hours thereafter up to hour 24 h, and then every 8 h up to 6 hour after the last ibuprofen dose.
Secondary efficacy endpoints | From 0 hours to 72 hours post- surgery
  - Ramsay-Hunt sedation scale.
Secondary efficacy endpoints | From 0 hours to 72 hours post- surgery
  - Time to first subsequent narcotic analgesia (or time to treatment failure).
Secondary efficacy endpoints | From 0 hours to 72 hours post- surgery
  - Number of doses of morphine and number of attempts of dosing at PCA
Secondary tolerability and safety endpoints | From 0 hours to 72 hours post- surgery
  - Report of adverse events (AEs) during the study
Secondary tolerability and safety endpoints | From 0 hours to 72 hours post- surgery
  - Local reactions due to IV infusion (pain, erythema, phlebitis)
Secondary tolerability and safety endpoints | From 0 hours to 72 hours post- surgery
  - Vital signs (heart rate, blood pressure, temperature) at 1, 3, 6 hour after the initial dose and every 8 hours thereafter.
Secondary tolerability and safety endpoints | From 0 hours to 72 hours post- surgery
  - Routine laboratory tests (chemistry, haematology and coagulation) at baseline and within 24 hours after the last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Concepción Pérez, MD, Study Chair — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa; Francisco Abad, MD, Study Chair — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa; Dolores Ochoa, MD, Study Chair — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa; Antonio Planas, MD, Study Chair — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (13):
- Spain (13):
  - Complejo Hospitalario Universitario de A Coruña, A Coruña, La Coruña
  - Hospital Arnau de Vilanova de Lleida, Lleida, Lleida
  - Hospital La Princesa, Madrid, Madrid
  - Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital de Montepríncipe, Madrid, Madrid
  - Hospital de Móstoles, Móstoles, Madrid
  - Clínica Universitaria de Navarra, Pamplona, Pamplona
  - Hospital Xeral Cíes de Vigo, Vigo, Pontevedra
  - Hospital Virgen de la Salud, Toledo, Toledo
  - Hospital La Fe, Valencia, Valencia
  - Hospital Clínico de Valladolid, Valladolid, Valladolid
  - Hospital de Cruces, Barakaldo, Vizcaya